CLINICAL TRIAL: NCT00709553
Title: A Randomised, Open-label, Crossover, Phase I Study to Assess the Effect of Multiple Oral Doses of ZD4054 (Zibotentan) on the Pharmacokinetics of a CYP450 3A Probe (Midazolam) in Healthy Male Subjects
Brief Title: Drug Interaction Study to Asses Multiple Doses of ZD4054 (Zibotentan)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Thomas Morris, BSc MB BCh MRCP FFPM, Medical Science Director, ZD4054, AstraZeneca R&D Alderley Park
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4320C00010; ZD4054EudraCt 2008-002764-35
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: ZD4054; Healthy Volunteers
MeSH Terms: interventions — Midazolam; ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): midazolam, one single dose of 705mg
  Interventions: Drug: midazolam
- 2 (Experimental): ZD4054(Zibotentan)- 10mg od, 7 days + midazolam (one single dose of 7.5 mg on day 6 )
  Interventions: Drug: midazolam; Drug: ZD4054

INTERVENTIONS:
Drug: midazolam
  Other Names: Dormicum®
Drug: ZD4054 — ZD4054 10 mg od
  Other Names: Zibotentan
  Arms: 2

SUMMARY:
The purpose of the study is to to assess the effect of multiple oral doses of ZD4054 (Zibotentan) on the pharmacokinetics of a CYP450 3A Probe (midazolam) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30 kg/m2
* Medical and surgical history and physical examination without any clinically significant findings
* Normal resting ECG with QTcB interval <450ms

Exclusion Criteria:

* Definite or suspected personal history or family history of hypersensitivity to drugs that are endothelin antagonists; ie, ambrisentan, artrasentan, sitaxsetan and bosentan
* Healthy volunteer has a known hypersensitivity to midazolam or any of the excipients of the midazolam tablet
* Medical diagnosis of migraine with an attack during the 12 months prior to Screening

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study

SECONDARY OUTCOMES:
Safety variables (adverse events, ECG, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morris, Study Director — AstraZeneca, Medical Science Director; Dago Mazur, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Derived] Tomkinson HK, Kemp JV, Wollseifen T, Morris T, Oliver SD. An open-label, randomized, single-center, two-period, phase I, crossover study of the effect of zibotentan (ZD4054) on the pharmacokinetics of midazolam in healthy male volunteers. Clin Ther. 2010 Jul;32(7):1372-86. doi: 10.1016/j.clinthera.2010.07.013. PMID 20678684